CLINICAL TRIAL: NCT05568589
Title: The Effects of Intraoperative and Preoperative Interpectoral -Pectoserratus Plan Block on Postoperative Pain, Amount of Analgesic Use, and Shoulder Joint Range of Motion in Patients Who Had Breast Cancer Surgery
Brief Title: Effects of Interpectoral-Pectoserratus Plane Block After Breast Cancer Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Izmir Bakircay University (Other)
Responsible Party: Principal Investigator, Omer Faruk Altas, Specialist, Izmir Bakircay University
Other Study IDs: 712
Record Dates: First submitted 2022-10-02; First posted 2022-10-05 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Pain, Postoperative; Disability Physical; Quality of Life
Keywords: İnterpectoral plane block; Pectoserratus plane block; Breast Cancer; PECS II Block
MeSH Terms: conditions — Pain, Postoperative; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Preoperative Interpectoral - Pectoserratus Plane Block: The block will be done by the Anesthesiologist.
  Interventions: Other: Preoperative Interpectoral - Pectoserratus Plane Block
- Intraoperative Interpectoral - Pectoserratus Plane Block: The block will be made by the surgeon.
  Interventions: Other: Intraoperative Interpectoral - Pectoserratus Plane Block
- Non Block: will not be blocked.
  Interventions: Other: Non Block

INTERVENTIONS:
Other: Preoperative Interpectoral - Pectoserratus Plane Block — Pain numerical rating scale (numering Rating Scale) at postoperative 1st, 2nd, 6th, 12th and 24th hours in patients, patient recovery scores at 24th hour (QoR15 Turkish version), amount of tramadol used in patient-controlled analgesia, time to first rescue analgesia , adverse events (pneumothorax, nausea, vomiting, pruritus, hematoma, allergic reactions) and hand grip strength on the postoperative 1st day, quality of life, shoulder joint range of motion, and disability level will be measured on the postoperative 10th day.
  Groups: Preoperative Interpectoral - Pectoserratus Plane Block
Other: Intraoperative Interpectoral - Pectoserratus Plane Block — Pain numerical rating scale (numering Rating Scale) at postoperative 1st, 2nd, 6th, 12th and 24th hours in patients, patient recovery scores at 24th hour (QoR15 Turkish version), amount of tramadol used in patient-controlled analgesia, time to first rescue analgesia , adverse events (pneumothorax, nausea, vomiting, pruritus, hematoma, allergic reactions) and hand grip strength on the postoperative 1st day, quality of life, shoulder joint range of motion, and disability level will be measured on the postoperative 10th day.
  Groups: Intraoperative Interpectoral - Pectoserratus Plane Block
Other: Non Block — Pain numerical rating scale (numering Rating Scale) at postoperative 1st, 2nd, 6th, 12th and 24th hours in patients, patient recovery scores at 24th hour (QoR15 Turkish version), amount of tramadol used in patient-controlled analgesia, time to first rescue analgesia , adverse events (pneumothorax, nausea, vomiting, pruritus, hematoma, allergic reactions) and hand grip strength on the postoperative 1st day, quality of life, shoulder joint range of motion, and disability level will be measured on the postoperative 10th day.
  Groups: Non Block

SUMMARY:
The aim of this study: It was aimed to observe the effects of intraoperative and preoperative PECS II block on postoperative pain, amount of analgesic use and shoulder joint range of motion in patients who underwent breast cancer surgery.

This research was planned as an observational study. For this purpose, patients who underwent breast cancer surgery in İzmir Bakırçay University Çiğli Training and Research Hospital General Surgery Clinic will be included in the study at the 1st hour after the operation. Patients who underwent preoperative Interpectoral - Pectoserratus Plan Block in the operation will be included in Group 1, patients who have been applied Interpectoral - Pectoserratus Plan Block between the muscle planes by the intraoperative surgeon will be included in Group 2, and patients who have not applied any block will be included in Group 3. Pain numerical rating scale (numering Rating Scale) at postoperative 1st, 2nd, 6th, 12th and 24th hours in patients, patient recovery scores (QoR15 Turkish version), amount of tramadol used in patient-controlled analgesia, time to first rescue analgesia, adverse events (pneumothorax, nausea, vomiting, itching, hematoma, allergic reactions) and quality of life, shoulder joint range of motion, hand grip strength (also on day 1) and disability level will be measured on postoperative day 10.

H0- Preoperative interpectoral - pectoserratus plane block affects the level of postoperative pain.

H1- Preoperativeinterpectoral - pectoserratus plane block does not affect the level of postoperative pain.

H2- Intraoperative interpectoral - pectoserratus plane block affects postoperative pain level H3- Intraoperative interpectoral - pectoserratus plane blockk does not affect the level of postoperative pain.

DETAILED DESCRIPTION:
Breast cancer is the most common type of cancer among women and the most common cause of death worldwide. While there has been a serious decrease in the mortality rate due to developments in diagnosis and treatment, there have been serious increases in functional disability and disability due to the disease. Breast cancer can lead to various functional losses due to the nature of the disease itself, radical surgical interventions and radiotherapy applications. These include shoulder dysfunction (pain and limitation of joint movement), locomotor system disorders such as upper extremity muscle strength loss and lymphedema, as well as psychological and cosmetic problems, and as a result, these problems affect the quality of life (QOL) of individuals (1).

Firstly, Blanco et al. Ultrasound-guided pectoralis nerve II block (Interpectoral and pectoserratus plan block - PECS II block), described by MD, is increasingly used for analgesia in breast surgery (2). It has been reported that PECS II block is effective in reducing postoperative pain intensity and opioid consumption (3). It is safe and relatively simple to apply as an interfascial plane block, and there is no sympathetic blockade (4). The PECS II block consists of two interfascial injections of local anesthetics: 1) between the pectoralis minor and serratus anterior muscles, 2) between the pectoralis major and pectoralis minor muscles at the level of the third rib. Local anesthetic injection into these planes; It is expected to block the lateral pectoral nerve, medial pectoral nerve, anterior branches of the thoracic intercostal nerves, and long thoracic nerves (5). Recently, the types of local anesthesia used during radical surgery may decrease the postoperative pain levels and recovery times of the patients. The effect of these intraoperative or postoperative blocks on the patients' clinical status in the postoperative period has not been compared before.

ELIGIBILITY:
Inclusion Criteria:

* Having had a unilateral breast cancer operation
* Signing the voluntary consent form

Exclusion Criteria:

* BMI >35kg/m2 and <20kg/m2
* Having a rheumatological disease (rheumatoid arthritis, etc.),
* Having neuromuscular disease
* Having a disease that will add shoulder joint movement (arthritis, prosthesis, fracture sequela, etc.)
* Having neuropathy, alcoholism, psychiatric disorder
* Chronic opioid use
* being pregnant
* Patient's refusal to use patient-controlled analgesia
* History of uncontrolled hypertension, diabetes, heart failure, liver failure, kidney failure and/or cerebrovascular disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sixty patients aged >18 years old who has breast cancer surgery with intraoperative or preoperative interpectoral - pectoserratus plane block o non block will be included in the study. Patients will be randomly divided into three groups including 20 patients each, postoperative 1st hour.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-10-06 (Estimated); Primary Completion 2023-01-06 (Estimated); Study Completion 2023-04-06 (Estimated)

PRIMARY OUTCOMES:
Postoperative opioid consumption | 24 hours
  Tramadol consumption in the first 24 hours after surgery

SECONDARY OUTCOMES:
NRS scores | 1., 2., 6., 12., 24. hour
  NRS scores in the first 24 hours after surgery
Quality of Recovery | 24th hours
  QoR-15 questionairre QoR-15 questionairre
The disability levels of the patients due to shoulder dysfunction. | 10th day
  The Shoulder Pain and Disability Index questionnaire will be used to determine The disability levels of the patients due to shoulder dysfunction. (Quick dash)
Hand grip muscle strength. | 24th hour, 10th day
  Hand grip muscle strength will be measured with a handheld dynamometer.
Quality of Life (Short Form 36) | 24th hour, 10th day
  The SF-36 Quality of Life scale will be used to assess quality of life.
Shoulder joint range of motion | 10th day
  Shoulder joint range of motion will be measured with a goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: Ömer Faruk Altaş, 1, Principal Investigator — İzmir Bakircay University
Locations (1):
- Izmir Bakircay University Cigli Training and Research Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No